CLINICAL TRIAL: NCT01787149
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicentre, Phase III Study to Evaluate the Efficacy and Safety of ENIA11 in Combination With DMARDs Versus DMARDs Alone in Patients With Rheumatoid Arthritis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mycenax Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TSHEN1201
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Combination With DMARDs
Keywords: ENIA11; DMARDs; RA; TNF
MeSH Terms: interventions — Antirheumatic Agents

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): DMARDs alone
  Interventions: Drug: DMARDs
- ENIA11 (Experimental): ENIA11 25 mg
  Interventions: Drug: DMARDs

INTERVENTIONS:
Drug: DMARDs

SUMMARY:
A Prospective, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicentre, Phase III Study to Evaluate the Efficacy and Safety of ENIA11 in Combination with DMARDs versus DMARDs Alone in Patients with Rheumatoid Arthritis

DETAILED DESCRIPTION:
The objectives of the study are to evaluate the efficacy and safety of ENIA11 in combination with DMARDs versus DMARDs alone in patients with rheumatoid arthritis.

This is a multi-center, double-blind, randomized, parallel-group, placebo-controlled study to evaluate the efficacy and safety of ENIA11 in combination with DMARDs versus DMARDs alone in patients with rheumatoid arthritis.

The study period for each patient will be 28 weeks, during which the patient will undergo screening for up to 14 days, followed by treatment of 24 weeks and follow-up period of 2 weeks. Each patient will be required to make a total of 9 visits.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥ 20 years old;
2. Patient meet ACR criteria for rheumatoid arthritis over 6 month duration;
3. Patient with active disease at the time of screening as defined by six or more swollen joints and six or more tender joints;
4. Presence of at least one of the following criteria:

   * Erythrocyte Sedimentation Rate (ESR) ≥ 28 mm/h,
   * C-Reactive Protein (CRP) ≥ 10 mg/L,
5. RA functional class I, II, or III;
6. Patients have been received stable doses of permitted DMARDs (methotrexate, hydroxychloroquine, sulfasalazine, azathioprine, and leflunomide) for at least 8 weeks prior enrollment.
7. Patient is willing and able to comply with study procedures and sign informed consent.

Exclusion Criteria:

1. Active autoimmune disease (other than RA) requiring immunosuppressive therapy;
2. In the opinion of the investigator, the patient shows persistent signs of immunosuppression;
3. Known hypersensitivity to etanercept or ENIA11 or any of its components;
4. Previous unsuccessful treatment with etanercept, anti-TNF monoclonal antibodies or a soluble TNF receptor (e.g., infliximab);
5. Suspected or diagnosed pulmonary tuberculosis, or other chronic or current infectious disease at discretion of investigator;
6. Patients who have a history or evidence of a medical condition that would expose them to an undue risk of a significant adverse event during the course of the trial, including but not limited to hepatic, renal, respiratory, cardiovascular, endocrine, immune, neurological, hematological, gastrointestinal or psychiatric disease as determined by the clinical judgment of the investigator;
7. Patients with any of the following laboratory abnormalities: ALT/AST > 3 times ULN, creatinine > 2 mg/dl, WBC < 3,000/mm3, Hgb < 8.5 g/dL, platelet count < 100,000/mm3;
8. Patients have received live attenuated vaccination program within 3 months or BCG vaccine within 12 months prior enrollment;
9. Female patient of childbearing potential who:

   * is lactating; or
   * has positive urine pregnancy test at Visit 1; or
   * refuse to adopt reliable method of contraception during the study;
10. Diagnosis of primary fibromyalgia or other joint inflammatory disease including but not limited to gout, reactive arthritis, psoriatic arthritis, seronegative spondyloarthropathy, Lyme disease;
11. Known or suspected positive serology for human immunodeficiency, hepatitis B or C virus;
12. Patient has received any investigational agent within 28 days or 5 half-lives, whichever is longer, prior to the first dose of investigational product;
13. Patient has history of substance abuse, drug addiction or alcoholism;
14. Patient who have had participated in prior phase I/II clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2013-09; Primary Completion 2017-12 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
ACR20 responder at last treatment visit | Week 24
  The primary efficacy endpoint is defined as ACR20 responder at last treatment visit (Week 24).

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao-Yi Lin, PHD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (7):
- Taiwan (7):
  - Cathay General Hospital, Taipei
  - Cheng Hsin General Hospital, Taipei
  - Far Eastern Memorial Hospital, Taipei
  - Mackay Memorial Hospital Institutional, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei City Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei